CLINICAL TRIAL: NCT07117331
Title: Efficacy of a Technology-Enhanced Continuous Nursing Intervention on Clinical Outcomes and Quality of Life Following Coronary Artery Bypass Grafting: A Randomized Controlled Trial
Brief Title: Technology-Enhanced Continuous Nursing System (TECNS) for Post-CABG Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Beibei Xing, Principal investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017S00298
Record Dates: First submitted 2025-07-30; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Technology-Enhanced Continuous Nursing System (TECNS) Group (Experimental): Patients received a comprehensive, 6-month continuous nursing program post-discharge. This included training on a dedicated smartphone app for educational modules; access to a moderated WeChat group for peer support and health tips; scheduled tele-rehabilitation calls from cardiac nurses for monitoring, education, and personalized guidance; and coordination with community health centers for follow-up. This was in addition to standard in-hospital care.
  Interventions: Behavioral: Technology-Enhanced Continuous Nursing System
- Active Comparator: Routine Care Group (Active Comparator): Patients received standard institutional postoperative care, including basic discharge education (oral and written summaries on medication, diet, and activity). Post-discharge care consisted of scheduled outpatient follow-up visits at 1 and 3 months post-surgery, without the technology-enhanced continuous support components.
  Interventions: Behavioral: Routine Postoperative Care

INTERVENTIONS:
Behavioral: Technology-Enhanced Continuous Nursing System — A multi-faceted behavioral and educational intervention lasting 6 months post-discharge. It utilized a smartphone app, WeChat, tele-monitoring (phone/video calls), and community health partnerships to provide structured education, personalized rehabilitation plans, and continuous professional nursing support.
  Arms: Experimental: Technology-Enhanced Continuous Nursing System (TECNS) Group
Behavioral: Routine Postoperative Care — Standard institutional care including standard discharge instructions and routine outpatient follow-up appointments.
  Arms: Active Comparator: Routine Care Group

SUMMARY:
This is a prospective, randomized controlled trial to evaluate the effectiveness of a Technology-Enhanced Continuous Nursing System (TECNS) compared to routine care for patients after coronary artery bypass grafting (CABG). The study aims to determine if the TECNS intervention, which includes digital health tools, personalized tele-rehabilitation, and continuous nursing support, can improve clinical outcomes such as postoperative hemoglobin recovery, reduce long-term major adverse cardiac events (MACE), and enhance patients' quality of life and psychological well-being.

DETAILED DESCRIPTION:
Patients undergoing coronary artery bypass grafting (CABG) face significant challenges during the post-discharge recovery period. The transition from hospital to home often creates a "care gap," where insufficient support and follow-up can lead to suboptimal outcomes, including poor medication adherence, increased complication rates, and diminished quality of life. This study was designed to address this gap by implementing and evaluating a Technology-Enhanced Continuous Nursing System (TECNS). Participants were randomized to receive either the comprehensive TECNS intervention for 6 months post-discharge or standard routine care. The TECNS intervention integrated a dedicated smartphone application for education, a WeChat group for peer and professional support, personalized tele-rehabilitation plans delivered by nurses, and coordination with community health centers. The study hypothesized that this proactive, continuous care model would lead to superior physiological recovery, better long-term clinical outcomes, and improved patient-reported outcomes compared to the traditional, fragmented approach to post-discharge care.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* Meeting diagnostic criteria for elective CABG
* Able to provide informed consent
* Owned a smartphone and was willing to use it for the study intervention

Exclusion Criteria:

* Emergency or salvage CABG
* Severe coexisting conditions that could confound outcomes (e.g., end-stage renal disease, severe COPD [GOLD stage IV], active malignancy)
* Left ventricular ejection fraction < 30%
* Participation in other clinical trials
* Severe cognitive impairment or psychiatric disorders precluding informed consent or adherence to the protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin (Hb) Level | Baseline, Day 7
  Change in blood hemoglobin concentration from baseline to 7 days after surgery, measured by laboratory analysis. This assesses the rate of postoperative hematopoietic recovery.
Major Adverse Cardiac Events (MACE)-Free Survival | Up to 24 months
  The rate of survival free from MACE, defined as a composite of cardiovascular death, non-fatal myocardial infarction, stroke, or unplanned revascularization.

SECONDARY OUTCOMES:
Change in Red Blood Cell Indices | Baseline, Day 7
  Change in Mean Corpuscular Volume (MCV), Red Blood Cell Distribution Width (RDW), and Hematocrit (HCT) from baseline.
Change in Quality of Life (QoL) | Baseline, 1 month, 3 months, 6 months
  Change in patient-reported quality of life assessed using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) scale. The scale ranges from 0 to 100. Higher scores indicate better QoL.
Patient Satisfaction | 1 month
  Patient-reported satisfaction with nursing care, assessed using a study-specific questionnaire. Responses are categorized ('Very Satisfied', 'Satisfied', 'Average', 'Dissatisfied').
Change in Interleukin-2 (IL-2) Level | Baseline, Day 7
  Change in serum level of Interleukin-2 (IL-2) from baseline, measured by laboratory analysis.
Change in Interleukin-6 (IL-6) Level | Baseline, Day 7
  Change in serum level of Interleukin-6 (IL-6) from baseline, measured by laboratory analysis.
Change in high-sensitivity C-reactive protein (hs-CRP) Level | Baseline, Day 7
  Change in serum level of high-sensitivity C-reactive protein (hs-CRP) from baseline, measured by laboratory analysis.
Change in Anxiety Symptoms | Baseline, 1 month, 3 months, 6 months
  Change in symptoms of anxiety assessed using the Self-Rating Anxiety Scale (SAS). The scale range is 25-100. Lower scores indicate better mental health (less anxiety).
Change in Depression Symptoms | Baseline, 1 month, 3 months, 6 months
  Change in symptoms of depression assessed using the Center for Epidemiologic Studies Depression Scale (CES-D). The scale range is 0-60. Lower scores indicate better mental health (less depression).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China